Cardiac surgery is associated with significant acute pain and a proportion of these patients will develop chronic post sternotomy pain (Ref 1, 2)

Opioids are the main stay of analgesia in cardiac surgery because of the safer hemodynamic profile and sedation (3). However high dose narcotic use is associated with a variety of unwanted side effects prolonging postoperative recovery. There is growing evidence for the effectiveness of multimodal approach utilizing opiate sparing techniques for enhancing patient recovery following surgery (4, 5, 6, 7). Early extubation has been associated with improved patient outcome and cost effectiveness in cardiac surgery (8, 9, 10).

Our objective is to assess the effectiveness of an opioid sparing multimodal approach for enhancing the recovery in Cardiac Surgical patients. This model would use a combination of intravenous (Dexmedetomidine, Ketamine, Lidocaine) and Intrathecal (Morphine) drugs.

All of the above anesthetic drugs have opioid sparing effect in surgical patients (11, 12,13).

Dexmedetomidine use has been associated with decreased atrial arrhythmias and improved neurological outcome in cardiac surgical patients (14, 15). Ketamine has been linked with attenuation of postoperative cognitive dysfunction after cardiac surgery (16,17).

Both intravenous lidocaine and intrathecal morphine has been shown to reduce narcotic consumption in the perioperative period (18, 19, 20)

## **Hypotheses**

Primary hypothesis – multimodal analgesia would improve pain scores at 24hr post extubation

Secondary hypothesis – multimodal approach would decrease opioid requirement in the first 24 hrs and enhance organ function recovery in the postoperative period

#### Methods:

Assuming mean pain score = 5 in control (21); test = 3 (2 point difference); stdev=2.5; n = 26/group (56 total subjects assuming a 8% drop out rate).

Prospective randomized trial with blinding at the stage of data analysis.

Study group: will receive pre-operative intrathecal duramorph (4mcg/kg up to max dose of 300mcg), intra-operative infusion of Ketamine (0.4 mg/kg/hr), Lidocaine (20 mcg/kg/min) and Dexmedetomidine (0.25 mcg/kg/hr) started after induction and maintained through the CPB towards the end of surgery. At this point all infusions will be turned off except Dexmedetomidine (0.25 mcg/kg/hr) which will be continued until the patient is extubated. The total intraoperative fentanyl dose will be limited to <250mcg (or 3mcg/kg). Control group: will receive unrestricted amount of intraoperative opioids at the discretion of the Anesthesiologist

Both groups will receive volatile agents and single dose of iv Tylenol intraoperatively and total midazolam to <2mg.

Postoperatively both groups will receive PRN iv Tylenol and PRN iv Opioids.

Inclusion criteria: Elective CABGs and/or Valve replacements

Exclusion criteria: Re-do cardiac surgery, Acute endocarditis, Circulatory arrest, Emergent cases, Shock, LVADs, Transplantation, TAVR, contraindications for neuraxial including coagulopathy and Clopidogrel <7days, psychosis, known allergy to any of the study drugs, Preoperative liver dysfunction (AST/ALT > 2 times normal) and Renal dysfunction (Cr > 2 mg/dL)

Drop outs: If a patient in the study group appears to require more narcotics than 250mcg of Fentanyl or midazolam >2mg, the patient will receive so and be dropped from the trial. Circumstances where the study protocol is not followed will lead to dropping out of those patients from the trial.

### **Outcome Measures**

Primary outcomes - Pain score at 24hr after extubation Secondary outcomes - Postoperative opioid consumption (in first 24 hrs), Extubation time, ICU Length of stay, Delirium scores, Inotropic requirement, patient satisfaction scores (in first 24 hrs)

#### **Data collection**

(Post op - Pain scores, sedation, nausea, vomiting, itching, hemodynamics, and respiratory parameters will be measured at 2, 4, 8, 12, 24, 48 & 72 hrs post extubation)

*Pain scores* – starting from 2hr post extubation, 11 point verbal rating scale, timing as above

*Opioid consumption* – first 12 hrs, thereafter daily and total (iv and PO)

Time of Extubation

*Lengths of stay*: ICU LOS, In-hospital LOS, 30 day readmission rate

Delirium: CAM-ICU measured at 24, 48 and 72 hrs

Inotrope requirement – Intraop, postoperative, total

*Patient satisfaction with pain management score*: in the first 24 hrs measured at above intervals

# **Complications**:

Cardiac complications: Atrial fibrillation on EKG, Arrhythmias requiring treatment, CHF (requiring 2 or more inotropes or use of IABP >24 hrs), MI (new Q waves in EKG or elevation of Troponins)

*Respiratory complications* – Mechanical ventilation >24hrs, desaturations, reintubations

*Neurological complications* – CVA, TIA, Post-operative delirium (measured by Delirium scores: CAM-ICU)

*Renal complications*: acute increase in Creatinine >50% of baseline or the need for dialysis

*Gastrointestinal complications*: Ileus (Measured as time of return of bowel function - POD to first oral liquid/flatus/stool)

*Infectious complications*: Surgical site infections, other organ infection, sepsis

*Opioid related Side effects*: Nausea, vomiting, pruritus, sedation (RASS score), urinary retention – measured as above

Other Perioperative and postoperative data collected: Anesthesia time, CPB time, Cross clamp time, Fluids, PRBC, FFP, Platelets, Cryoppt, Urine output, Electrical defibrillation, No of defibrillations, Pacing, Time of ventilation weaning

#### **References:**

- **1.** Lahtinen P, Kokki H, Hynynen M: Pain after cardiac surgery: A prospective cohort study of 1-year incidence and intensity. Anesth esiology 2006; 105:794–800
- 2. Choinie` re M, Watt-Watson J, Taillefer M, et al. Prevalence of and risk factors for persistent postoperative nonanginal pain after cardiac surgery: a 2-year prospective multicentre study. Can Med Assoc J 2014; 186:E213–E233
- 3. Lowenstein E, Hallowell P, Levine FH, Daggett WM, Austen WG, Laver MB. Cardiovascular response to large doses of intravenous morphine in man. N Engl J Med 1969;281:1389–93
- **4.** Kehlet H, Dahl JB: The value of "multimodal" or "balanced analgesia" in post-operative pain treatment. Anesth Analg 1993; 77:1048–56
- **5.** Varadhan KK, Neal KR, Dejong CH, Fearon KC, Ljungqvist O,Lobo DN. The enhanced recovery after surgery (ERAS) pathway for patients undergoing major elective open colorectal surgery: a meta-analysis of randomized controlled trials. Clin Nutr 2010;29:434–40

- 6. Marret E, Remy C, Bonnet F; Postoperative Pain Forum Group. Metaanalysis of epidural analgesia versus parenteral opioid analgesia after colorectal surgery. Br J Surg 2007;94:665–73
- <u>7.</u> Junger A, Klasen J, Benson M, et al. Factors determining length of stay of surgical day-case patients. Eur J Anaesthesiol 2001;18:314-21
- **8.** Hawkes, C. A., S. Dhileepan, and D. Foxcroft. "Early Extubation for Adult Cardiac Surgical Patients." The Cochrane database of systematic reviews (4).4 (2003): CD003587
- **9.** Zhu, F., A. Lee, and Y. E. Chee. "Fast-Track Cardiac Care for Adult Cardiac Surgical Patients." The Cochrane database of systematic reviews 10 (2012): CD003587
- **10.** Myles, P. S., and D. McIlroy. "Fast-Track Cardiac Anesthesia: Choice of Anesthetic Agents and Techniques." Seminars in cardiothoracic and vascular anesthesia 9.1 (2005): 5-16
- **11.** De Oliveira GS Jr, Fitzgerald P, Streicher LF, et al. Systemic lidocaine to improve postoperative quality of recovery after ambulatory laparoscopic surgery. Anesth Analg 2012;115:262-7
- **12.** Loftus RW, Yeager MP, Clark JA, et al. Intraoperative ketamine reduces perioperative opiate consumption in opiate-dependent patients with chronic back pain undergoing back surgery. *Anesthesiology* 2010;113:639–646
- **13.** Tan JA, Ho KM. Use of dexmedetomidine as a sedative and analgesic agent in critically ill adult patients: a meta-analysis. Intensive Care Med 2010; 36:926–939
- **14.** Turan A, Bashour CA, You J, Kirkova Y, Kurz A, Sessler DI and Saager L: Dexmedetomidine sedation after cardiac surgery decreases atrial arrhythmias. J Clin Anesth 26: 634-642, 2014
- **15.** Ji, F., Li, Z., Nguyen, H., Young, N., Shi, P., Fleming, N., & Liu, H. (2013). Perioperative dexmedetomidine improves outcomes of cardiac surgery. *Circulation*, CIRCULATIONAHA-112
- **16.** Hudetz JA, Iqbal Z, Gandhi SD *et al.* Ketamine attenuates post-operative cognitive dysfunction after cardiac surgery. Acta Anaesthesiol Scand 2009;53:864–7
- **17.** Botero C, Smith C, Holbrook C, et al. Total intravenous anesthesia with a propofol-ketamine combination during coronary artery surgery. J Cardiothorac Vasc Anesth 2000;14:409–15
- **18.** Insler, SR, O'Connor, M, Samonte, AF (1995) Lidocaine and the inhibition of postoperative pain in coronary artery bypass patients. J Cardiothorac Vasc Anesth 9: pp. 541-6
- **19.** Chaney MA. Intrathecal and epidural anesthesia and analgesia for cardiac surgery. Anesth Analg.2006;102:45–64
- **20.** Chaney MA, Smith KR, Barclay JC, Slogoff S. Large-dose intrathecal morphine for coronary artery bypass grafting. Anesthesia and analgesia. 1996;83:215–22
- **21.** Murphy GS, Szokol JW, Marymont JH, et al. Morphine based cardiac anesthesia provides superior early recovery compared with fentanyl in elective cardiac surgery patients. Anesth Analg 2009; 109:311–9